CLINICAL TRIAL: NCT03303885
Title: The FGF/FGFR Signalling Pathway: a Novel Therapeutic Target in Liposarcomas
Brief Title: The FGF/FGFR Signalling Pathway:
Acronym: FILIPO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 16-PRTK
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Liposarcoma
MeSH Terms: conditions — Liposarcoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Liposarcoma biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
Liposarcomas are the most common type of soft tissue sarcomas (STS). Among liposarcomas, well-differentiated liposarcoma (WDLPS)/dedifferentiated liposarcoma (DDLPS) are the most frequent types. WDLPS are composed mostly of mature fat whereas DDLPS contain both a WDLPS component and a non-lipomatous sarcoma component mostly of high grade. More than 50% of DDLPS will relapse locally. A significant proportion of patients will remain with a non-resectable disease that will metastasize in 20% of cases. Standard chemotherapy is poorly efficient and alternative options are so far limited. Identification of new therapeutic targets is urgent and mandatory. the recent preliminary results as well as data from the literature led us to hypothesize that the FGF (Fibroblast Growth factor)/FGFR pathway is involved in liposarcomagenesis and might therefore be a novel relevant therapeutic target in WDLPS/DDLPS.

Description of the project The project associates 4 teams with a longstanding collaboration : 3 teams fom Nice (Nice University Hospital/IRCAN, Nice University Hospital, Comprehensive Cancer Center Centre Antoine Lacassagne and one team from Bordeaux (Comprehensive Cancer Center Institut Bergonié). These 4 teams are experts in the clinics, pathology and molecular genetics of sarcomas as well as in biostatistics.

1. Expression studies on the role of the syndecan-1 (SDC1)/FGFR pathway in WDLPS/DDLPS tumorigenesis

   The recent studies provide original results that may have a direct application in treatments of liposarcomas. They suggest that SDC1 -an effector of the FGF/FGFR pathway- might be involved in DDLPS tumorigenesis. Staff will analyse:
   * The pattern of expression and localisation of syndecans, FGFs and FGFRs in WDLPS/DDLPS both in a large collection of 249 primary tumors and in our in-house panel of high quality and validated human WDLPS/DDLPS cell lines.
   * The prognostic value of SDC1, FGF2 and FGF18 expression by correlation to the patient clinical outcomes
2. Fonctional studies of the role of the SDC1/FGFR pathway in WDLPS/DDLPS tumorigenesis. We will analyse:

   * The effects of modulating SDC1, FGFR expression in WDLPS and DDLPS cells on cell proliferation, cell cycle, apoptosis and on their capacity to differentiate in adipocytes.
   * The sensitivity of WDLPS and DDLPS cells to the FGFR inhibitor JNJ-427556493 as a single agent or in combination with other antagonists.
   * The mechanisms of sensitivity and resistance to JNJ-427556493 by phosphoproteomic analysis of WDLPS and DDLPS cells before and after JNJ-427556493 treatment.
   * The involvement of SDC1 in the dedifferentiation process of liposarcoma. Expected results staff expect to demonstrate the relevance of the SDC1/FGFR pathway in liposarcomas. We also expect to link drug activity to genomics and proteomics data. This will allow the characterization of the activity of FGFR inhibitors and the identification of powerful preclinical biomarkers of drug activity and mechanisms of resistance in DDLPS. The availability of xenograft models will allow us to validate our in vitro findings in the in vivo setting with the ultimate goal to improve patient management.

The availability of an early clinical trial unit in Institut Bergonié, managed by A. Italiano, will give the immediate opportunity to transfer our data to the management of metastatic liposarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

* A biopsy and\or an exérèse with diagnostic or curative aim will have been practised within the framework of a well differentiated liposarcome or dédifférencié with development of the gene MDM2
* A taking of the tumor is available (frozen fragment and\or block fixed in paraffin wax) - not opposition of the patient will have been looked for

Exclusion Criteria:

Liposarcome not differentiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: biopsy of liposarcoma patient
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
difference in terms of overall survival: between FGF18 - versus FGF18+ | 24 months
  overall survival, recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided